CLINICAL TRIAL: NCT04202029
Title: Additional Benefit of Thoracic Impedance Monitoring (TIM) for Propofol-sedation Monitoring by Non- Anesthesiologist During Percutaneous Endoscopic Gastrostomy (PEG), a Prospective, Randomized-controlled Clinical Study.
Brief Title: Additional Benefit of Thoracic Impedance Monitoring (TIM) for Propofol-sedation Monitoring During PEG Placement
Acronym: TIMPEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georg Dultz (Other)
Responsible Party: Sponsor-Investigator, Georg Dultz, Clinical Professor, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FRA-UNI-TIM-PEG-TRIAL-2019
Record Dates: First submitted 2019-11-03; First posted 2019-12-17 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2020-05

CONDITIONS: Percutaneous Endoscopic Gastrostomy (PEG)
Keywords: ASA; American Socity of Anesthesiologists physical status classification system; Thoracic Impedance monitoring; TIM; ECG; echocardiography; sedation; propofol; monitoring; NAPS; nurse-administered propofol sedation; O2; oxygen; PEG; percutaneous endoscopic gastrostomy

STUDY DESIGN:
Intervention Model Description: The participants will be randomely assigend by a computer based algorithm to either the standard monitoring group as defined by the German S3 guidline "Sedierung in der gastrointestinalen Endoskopie" containing pulsoxymetry and non-invasive blood preassure monitoring versus the standard and additionally the thoracic impedance monitoring using an extra ECG
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulseoxymetry arm (Other): pulseoxymetry arm: standard monitoring: pulseoxymetry and non-invasive blood preassure monitoring
  Interventions: Device: pulseoxymetry; Device: non-invasive blood preassure monitoring
- thoracic impedance monitoring arm (Experimental): thoracic impedance monitoring arm: standard monitoring and additionally thoracic impedance measurement)
  Interventions: Device: thoracic impedance monitoring; Device: pulseoxymetry; Device: non-invasive blood preassure monitoring

INTERVENTIONS:
Device: thoracic impedance monitoring — Thoracic impedance measurement identifies the respiratory frequence using the changes of impedance during inspiration and expiration via an ECG.
  Arms: thoracic impedance monitoring arm
Device: pulseoxymetry — Pulseoxymetry is meassuring the heart rate and the oxygen saturation in the arterial blood
Device: non-invasive blood preassure monitoring — Non-invasive blood preassure is a method using a blood preassure cuff to identify the blood preassure.

SUMMARY:
The present study is a randomized, prospective, single-blinded study. A total of 172 patients presenting for percoutaneous endoscopic gastrostomy (PEG) under sedation will be included according to the statistical sample size calculation. Patients will be randomized to either group 1- standard monitoring (pulseoxymetry and non-invasive blood preassure monitoring) or group 2- standard monitoring and thoracic impedance measurement during Propofol-based sedation for PEG. Episodes of Hypoxia are documented and compared in both groups.

Statistical analysis will be done in cooperation with the statistical biomedical institute oft he university hospital in Frankfurt.

ELIGIBILITY:
Inclusion Criteria:

* > /= 18 years
* given consent
* planned PEG

Exclusion Criteria:

* ASA >/= 4
* no given consent
* pregnant/laction
* contraindication against PEG
* contraindication against propofol-sedatation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
comparison of hypoxia in both arms | Average duration period of PEG-placement: approx. 15 minutes.
  Hypoxia is defined as oxygen saturation dropping below 90 % for more than 15 seconds. The primary end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by awaking of the patient.

SECONDARY OUTCOMES:
Comparison of hypoxia-episodes in both arms | Average duration period of PEG-placement: approx. 15 minutes.
  Number of hypoxia-episodes during each intervention. This end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by awaking of the patient.
Comparison of severe hypoxia episodes in both arms defined as oxygen saturation dropping below 85 % | Average duration period of PEG-placement: approx. 15 minutes.
  Severe hypoxia is defined as O2 saturation below 85%. This end point is assessed from the beginning of propofol sedatio n until the PEG-procedure is terminated defined by awaking of the patient.
Comparison of severe hypoxia-episodes in both arms | Average duration period of PEG-placement: approx. 15 minutes. This end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by awaking of the patient.
  The number of hypoxia-episodes during each intervention will be assesed. This end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by awaking of the patient.
Comparison of the time difference of occuring apnoe before hypoxia | Average duration period of PEG-placement: approx. 15 minutes.
  The time difference between the onset of apnoe befpre the onset of hypoxia will be meassured.
Specifity and sensetivity of thoracic impedance monitoring | Average duration period of PEG-placement: approx. 15 minutes.
  The specifity and sensitivity will be calculated using the frequency of falls alarms and missed alarms in relation to hypoxia. This end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by awaking of the patient.
Additional cost of thoracic impedance monitoring (TIM) | Time frame is the entire study period with a maximum of 3 years.
  The costs that are needed to implement TIM during every procedure will be calculated and will be stated in the results. All PEG-placements in the TIM group will be used. By using a 3-lead-ECG, 3 electrodes will be needed per patient. For alle patients, one ECG-cable will be needed. Therefore, the costs will be calculated per patient.
Risk stratification of baseline criteria for hypoxia | Time frame is the entire study period with a maximum of 3 years.
  Risk factors will be evaluated in an univariate and a multivariate analyse
Comparison of intervention procedures to prevent hypoxia | Average duration period of PEG-placement: approx. 15 minutes.
  The necessity to prevent a hypoxic event because of an alarm by the monitoring by elevating the oxygen delivery, using jaw thrust manoeuvre or mask ventilation will be compared in both arms. This end point is assessed from the beginning of propofol sedation until the PEG-procedure is terminated defined by the awaking of the patient.
Comparison of satisfaction of doctors in both arms | approx. 15 minutes
  The involved doctors will be asked to give there opinion using visual analog scale (VAS). Scale reaches from 1 (dissatisfied) to 10 (satisfied). The end point will be meassured after the procedure. The investigation time is defined as one PEG-placement.
Comparison of satisfaction of nurses in both arms | approx. 15 minutes
  The involved nurses will be asked to give there opinion using visual analog scale (VAS). Scale reaches from 1 (dissatisfied) to 10 (satisfied). The end point will be meassured after the procedure. The investigation time is defined as one PEG-placement.
Comparison of satisfaction of patients in both arms | approx. 15 minutes
  The involved patients will be asked to give there opinion using visual analog scale (VAS). Scale reaches from 1 (dissatisfied) to 10 (satisfied). The end point will be meassured after the procedure. The investigation time is defined as one PEG-placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafari A, Weismuller TJ, Tonguc T, Kalff JC, Manekeller S. [Complications after Percutaneous Endoscopic Gastrostomy Tube Placement - A Retrospective Analysis]. Zentralbl Chir. 2016 Aug;141(4):442-5. doi: 10.1055/s-0035-1557765. Epub 2015 Aug 10. German. PMID 26258619
- [Background] Riphaus A, Rabofski M, Wehrmann T. Endoscopic sedation and monitoring practice in Germany: results from the first nationwide survey. Z Gastroenterol. 2010 Mar;48(3):392-7. doi: 10.1055/s-0028-1109765. Epub 2010 Feb 5. PMID 20140841
- [Background] Riphaus A, Geist F, Wehrmann T. Endoscopic sedation and monitoring practice in Germany: re-evaluation from the first nationwide survey 3 years after the implementation of an evidence and consent based national guideline. Z Gastroenterol. 2013 Sep;51(9):1082-8. doi: 10.1055/s-0033-1335104. Epub 2013 Sep 10. PMID 24022202
- [Background] Lin OS. Sedation for routine gastrointestinal endoscopic procedures: a review on efficacy, safety, efficiency, cost and satisfaction. Intest Res. 2017 Oct;15(4):456-466. doi: 10.5217/ir.2017.15.4.456. Epub 2017 Oct 23. PMID 29142513
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anaesthesiologist administration of propofol for GI endoscopy. Eur J Anaesthesiol. 2010 Dec;27(12):1016-30. doi: 10.1097/EJA.0b013e32834136bf. PMID 21068575
- [Background] Riphaus A, Wehrmann T, Hausmann J, Weber B, von Delius S, Jung M, Tonner P, Arnold J, Behrens A, Beilenhoff U, Bitter H, Domagk D, In der Smitten S, Kallinowski B, Meining A, Schaible A, Schilling D, Seifert H, Wappler F, Kopp I; German Society of General and Visceral Surgery; German Crohn's disease / ulcerative colitis Association e. V; German Society of Anaesthesiology and Intensive Care Medicine e. V. (DGAI); Gesellschaft Politics and Law in Health Care (GPRG). [S3-guidelines "sedation in gastrointestinal endoscopy" 2014 (AWMF register no. 021/014)]. Z Gastroenterol. 2015 Aug;53(8):802-42. doi: 10.1055/s-0035-1553458. Epub 2015 Aug 18. No abstract available. German. PMID 26284330
- [Background] Absolom M, Roberts R, Bahlmann UB, Hall JE, Armstrong T, Turley A. The use of impedance respirometry to confirm tracheal intubation in children. Anaesthesia. 2006 Dec;61(12):1145-8. doi: 10.1111/j.1365-2044.2006.04838.x. PMID 17090233
- [Background] Frasca D, Geraud L, Charriere JM, Debaene B, Mimoz O. Comparison of acoustic and impedance methods with mask capnometry to assess respiration rate in obese patients recovering from general anaesthesia. Anaesthesia. 2015 Jan;70(1):26-31. doi: 10.1111/anae.12799. Epub 2014 Jul 10. PMID 25040754